CLINICAL TRIAL: NCT03508973
Title: Sculptra for Décolletage Crepiness and Wrinkling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skin Laser & Surgery Specialists (Other)
Responsible Party: Principal Investigator, David J. Goldberg, MD, David J. Goldberg, MD, JD, Skin Laser & Surgery Specialists
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCULPTDEC01
Record Dates: First submitted 2016-05-26; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Décolletage

ARMS (1):
- Sculptra (Experimental): Sculptra, an injectable implant containing microparticles of ply-L-lactic acid, carboxymethylcellulose, non-pyrogenic mannitol and sterile water, will be injected into the decolletage.
  Interventions: Other: Sculpta

INTERVENTIONS:
Other: Sculpta

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Sculptra as a volume agent to improve décolletage crepiness and wrinkling.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteer
* Aged from 40-70 years on the day of screening
* No known medical conditions that may interfere with study participation
* Moderate to severe crepiness and wrinkling of the décolletage
* Willingness to not use any products on their décolleté for the duration of the study
* Read, understand, and sign informed consent forms
* Willingness to sign photography release form
* Willing and able to comply with all follow-up requirements
* Willingness to undergo a series of three Sculptra injections, 2-3 months apart, in their décolletage

Exclusion Criteria:

* Any significant skin disease at treatment area
* Any medical condition which could interfere with the treatment
* Inability or unwillingness to follow the treatment schedule
* Inability or unwillingness to sign the informed consent
* History of poor wound healing
* History of keloid formation
* History of HIV, hepatitis, immuno-compromised
* Pregnant or lactating
* Previous use of deep chemical peels on the treatment area
* Previous injections of Sculptra in the décolletage
* Known hypersensitivity to Sculptra or any of its ingredients
* Previous laser or light based treatments to the treatment area 6 months prior to the screening visit

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2016-12-13 (Actual)

PRIMARY OUTCOMES:
Change in décolletage crepiness and wrinkling in treatment area as measured by 5 point décolletage wrinkle scale | Screening, Treatment 1, Treatment 2, Treatment 3, 1 Month Follow up, 3 Month Follow up and 6 Month Follow up